CLINICAL TRIAL: NCT02136797
Title: A Phase II Trial of Third Party Donor Derived CMVpp65 Specific T-cells for The Treatment of CMV Infection or Persistent CMV Viremia After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Trial of Third Party Donor Derived CMVpp65 Specific T-cells for The Treatment of CMV Infection or Persistent CMV Viremia After Allogeneic Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-070
Expanded Access: NCT03010332 (No longer available)
Record Dates: First submitted 2014-05-09; First posted 2014-05-13 (Estimated); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-07

CONDITIONS: CMV Infection; Persistent CMV Viremia
Keywords: CMVpp65 Specific T-cells; Allogeneic Hematopoietic Stem Cell Transplantation; 14-070
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CMVpp65-CTL T-cells (Experimental): The T-cells to be infused will be selected from our bank of GMP grade CMVpp65-CTL. T-cells will be administered by bolus intravenous infusion. In this phase II trial, patients will be treated at doses of 1 x 10^6 CMVpp65-CTL/kg/dose/week for 3 weeks. Patients will be observed for the following 3 weeks. Additional 3 week courses of CMVpp65-CTL may be administered if levels of CMV DNA in blood are still detectable despite disease stabilization or improvement.
  Interventions: Biological: CMVpp65 Specific T-cells

INTERVENTIONS:
Biological: CMVpp65 Specific T-cells

SUMMARY:
The purpose of this study is to see how well transfusions of T-cells work in treating CMV. Tcells are a type of white blood cell that helps protect the body from infection. A transfusion is the process by which blood from one person is transferred to the blood of another. In this case, the T-cells are made from the blood of donors who are immune to CMV. The T-cells are then grown and taught to attack the CMV virus in a lab.

ELIGIBILITY:
Inclusion Criteria:

* Each patient must satisfy at least one of the following criteria:

  1. The patient must have a clinically documented condition associated with CMV (e.g. interstitial pneumonia, hepatitis, retinitis, colitis) Or
  2. The patient must have microbiological evidence of CMV viremia or tissue invasion as attested by viral culture, or detection of levels of CMV DNA in the blood or body fluids consistent with CMV infection.
* Patient must also satisfy at least one of the following criteria:

  1. The patient's CMV infection is clinically progressing or CMV viremia is persistent or increasing (as evidenced by quantitation of CMV DNA in the blood) despite two weeks induction therapy with antiviral drugs.

     Or
  2. The patient has developed CMV viremia as attested by viral culture, or detection of levels of CMV DNA in blood or body fluids while receiving prophylactic doses of antiviral drugs to prevent CMV infection post transplant.

     Or
  3. The patient is unable to sustain treatment with antiviral drugs due to drug associated toxicities (e.g. myelosuppression [ANC< 1000μl/ml without GCSF support] or nephrotoxicity [corrected creatinine clearance ≤ 60 ml/min/1.73 m^2 or serum creatinine > 2 mg/dl]) CMV infections are life threatening, and may involve multiple organ systems such as the lungs, liver, gastrointestinal tract, hematopoietic and central nervous systems. Antiviral drugs used for treatment may also compromise renal and hematopoietic function. Therefore, dysfunctions of these organs will not affect eligibility for this protocol.
* Patients must meet the following clinical criteria to receive CMVpp65-CTL infusions

  1. Stable blood pressure and circulation, not requiring pressor support
  2. Evidence of adequate cardiac function as demonstrated by EKG and/or echocardiography.
  3. A life expectancy of at least 3 weeks, even if requiring artificial ventilation.
  4. There are no age restrictions
* Patient must also satisfy at least one of the following criteria:

  1. The patient's HCT donor has not been previously infected by or sensitized to CMV (e.g. a cord blood transplant or a marrow or PBSC transplant from a seronegative donor).
  2. The patient's HCT donor, if seropositive, is either not available or not willing to provide leukocytes for generation of CMV-specific T-cells.
  3. There are CMVpp65-specific T-cells available in appropriate doses in the MSKCC Adoptive Immune T-cell Therapy Bank that are matched with the patient for 1 HLA allele and that exhibit CMVpp65-specific cytotoxic activity that is restricted by an HLA allele shared by the patient

Exclusion Criteria:

* Patients requiring high doses of glucocorticosteroids (≥ 0.3 mg/kg prednisone or its equivalent)
* Patients who are moribund
* Patients with other conditions not related to CMV infection (e.g. uncontrolled bacterial sepsis or invasive fungal infection) which are also life-threatening and which would preclude evaluation of the effects of a T-cell infusion.
* Patients who are pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-05-08 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Prockop, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- CMVpp65-CTL T-cells: The T-cells to be infused will be selected from our bank of GMP grade CMVpp65-CTL. T-cells will be administered by bolus intravenous infusion. In this phase II trial, patients will be treated at doses of 1 x 10^6 CMVpp65-CTL/kg/dose/week for 3 weeks. Patients will be observed for the following 3 weeks. Additional 3 week courses of CMVpp65-CTL may be administered if levels of CMV DNA in blood are still detectable despite disease stabilization or improvement.
  CMVpp65 Specific T-cells
Period: Overall Study
Arm/Group | CMVpp65-CTL T-cells
Started | 77
Completed | 69
Not Completed | 8
Not completed — Not Treated | 8

BASELINE CHARACTERISTICS:
Arm/Group | CMVpp65-CTL T-cells
Number analyzed (Participants) | 77
Age, Continuous [Median (Full Range); unit: years] | 43 [0 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 64
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 51
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 77

OUTCOME MEASURES:

1. Primary Outcome: Complete Response
Description: defined as the clearance of the CMV infection 3-7 weeks following completion of the last cycle of CMV CTLs.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | CMVpp65-CTL T-cells
Number analyzed (Participants) | 77
Participants
  Participants with Complete Response | 20
  Participants without Complete Response | 57

2. Secondary Outcome: Number of Participants With SAE's Possibly Related to Study Treatment
Description: Will be capturing and tracking Grade 3-5 toxicities which occur within 30 days following an infusion of CMVpp65-specific. For the evaluation of toxicities, the NCI Standard Toxicity Scale 4.0 will be employed.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | CMVpp65-CTL T-cells
Number analyzed (Participants) | 77
Participants
  Participants with possibly related SAE | 6
  Participants without possibly related SAE | 71

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | CMVpp65-CTL T-cells
All-Cause Mortality (participants affected / at risk) | 16/77
Serious Adverse Events (participants affected / at risk) | 22/77
Other Adverse Events (participants affected / at risk) | 9/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CMVpp65-CTL T-cells (N=77)
Acute coronary syndrome (Cardiac disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Autoimmune disorder (Immune system disorders) | 2
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 3
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Catheter related infection (Infections and infestations) | 4
Confusion (Psychiatric disorders) | 1
Death NOS (General disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Ejection fraction decreased (Investigations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Fever (General disorders) | 1
Headache (Nervous system disorders) | 1
Heart failure (Cardiac disorders) | 3
Hematuria (Renal and urinary disorders) | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Hypertension (Vascular disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypotension (Vascular disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Iron overload (Metabolism and nutrition disorders) | 1
Lung infection (Infections and infestations) | 3
Lymphocyte count decreased (Investigations) | 1
Multi-organ failure (General disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Neutrophil count decreased (Investigations) | 3
Pericardial effusion (Cardiac disorders) | 1
Platelet count decreased (Investigations) | 4
Resp, thoracic & mediastinal disorder Other, spec (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9
Retinal detachment (Eye disorders) | 1
Sepsis (Infections and infestations) | 4
Sinus bradycardia (Cardiac disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CMVpp65-CTL T-cells (N=77)
Blood and lymphatic system disorders - Other, spec (Blood and lymphatic system disorders) | 1
Encephalitis infection (Infections and infestations) | 1
Heart failure (Cardiac disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Lung infection (Infections and infestations) | 1
Pericardial effusion (Cardiac disorders) | 1
Platelet count decreased (Investigations) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/97/NCT02136797/Prot_SAP_000.pdf